CLINICAL TRIAL: NCT05554081
Title: Effect of Standardization of Urine Collection Using PEEZY Device as Compared to Clean Catch in the Detection of Asymptomatic Bacteriuria in an Obstetric Population
Brief Title: Effect of Standardization of Urine Collection Using PEEZY Device as Compared to Clean Peezy for DAB
Acronym: Peezy-DAB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, ann.lal, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 216104
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Asymptomatic Bacteriuria; Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Clean catch BMI < 30 (Placebo Comparator): Standard of care urine collection
  Interventions: Device: Peezy urine collection device
- Clean catch BMI > 30 (Placebo Comparator): Standard of care urine collection
  Interventions: Device: Peezy urine collection device
- PEEZy collection BMI < 30 (Experimental): PEEZY device for urine collection
  Interventions: Device: Peezy urine collection device
- PEEZY collection BMI > 30 (Experimental): PEEZY device for urine collection
  Interventions: Device: Peezy urine collection device

INTERVENTIONS:
Device: Peezy urine collection device — use peezy collection to obtain urine sample

SUMMARY:
This study aims specifically to compare the rates of contaminants between standard clean-catch urine collection and urine collected using the PEEZY device. In particular, this study will compare the rates of contamination as stratified by BMI status (i.e., BMI < 30 and BMI ≥30). Based on previous studies through LUHS and the Wolfe lab, we anticipate a reduction in contamination from sample collected using the PEEZY device, particularly among those pregnant women with BMI ≥30. To investigate this hypothesis we have designed a prospective unblinded randomized controlled trial comparing voided urine specimens obtained for asymptomatic bacteriuria in pregnant women presenting for obstetric care with use of standard clean-catch (CC) sampling method versus specimen obtained using PEEZY collection device.

DETAILED DESCRIPTION:
Recruitment procedures

1. All patients scheduled for "NOB" (new obstetrics) appointments at LOC will be screened for eligibility by residents and fellows
2. Residents and fellows will recruit participants at LOC and obtain informed consent.
3. There will not be any advertising for this study and no recruitment materials will be given to eligible participants.

   Study procedures
4. Residents and fellows will use a REDCaps database to assign randomization, generate de-identified study labels, and provide study participants with assigned urine collection device as well as instructions on use.
5. Participants will use a private bathroom to void and collect their urine specimen using either the PEEZY device or standard clean catch method as assigned.
6. Urine specimens will be handed to LOC nursing staff who will separate into 3 aliquots - 1 for clinical lab and 2 for Wolfe lab.
7. Wolfe lab aliquots will be labeled with the subject's study ID and placed at 4°C for <4 hours before transport to Dr. Wolfe's laboratory for inventory, storage and analysis
8. Clinical lab specimen will be labeled with patient label and transported to clinical lab for standard urine culture per routine obstetric care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant < 20 weeks gestational age
* Age > 18 years old
* English speaking

Exclusion Criteria:

* History of recurrent UTIs
* Need for ongoing antibiotics
* Urinary tract anomalies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Urine contamination rates | August 2022-August 2023
  1. To compare the rates of contaminants between CC and PEEZY samples stratified by BMI status (i.e., BMI < 30 and BMI ≥30)

SECONDARY OUTCOMES:
Maternal comorbidities and contamination | August 2022-August 2023
  To compare the rates of contamination based on maternal medical comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No